CLINICAL TRIAL: NCT00408941
Title: EEG and Auditory Evoked Potentials During Local Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1505/06
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-12

CONDITIONS: Healthy
Keywords: EEG; AEP; Artefacts; Propofol; Local Anaesthesia
MeSH Terms: interventions — Propofol; Prilocaine

INTERVENTIONS:
Drug: Propofol
Drug: Prilocaine

SUMMARY:
The aim of the present study was to investigate the sensitivity of AEP (auditory evoked potentials) to muscular artefacts using sedation and local anesthesia.

DETAILED DESCRIPTION:
Spontaneous or evoked electrical brain activity is increasingly used to monitor general anesthesia. During alertness, surgery and anesthesia the quality of AEP recordings may be reduced by artefacts. This poses the question to what extent AEP are sensitive for muscular artefacts. High frequency artefacts can have its seeds in muscles and in technical instruments in the operating room. Therefore, the study will take place under the terms of laboratory.

The present study was designed to measure the influence of muscular artefacts on AEP under propofol sedation with or without local anesthesia in the area of the electrodes.

If artefacts influence AEP, which are used to measure anesthesia, it is particularly interesting with regard to clinical application. AEP as a measure of "anesthetic depth" may not only reflect brain, but also muscular and high frequency activity. Therefore, while using muscle relaxants, the AEP of an awake patient may indicate deep anesthesia, because muscle signals are absent.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1-2

Exclusion Criteria:

* drugs that effect the central nervous system
* neurological or psychiatric deceases
* contraindications against use of propofol or local anesthesia

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15
Dates: Start 2006-12; Study Completion 2006-12

PRIMARY OUTCOMES:
differences of AEP during sedation with and without local anaesthesia

SECONDARY OUTCOMES:
fraction of high frequency artefacts
time to LOC
differences AEP awake with and without local anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Kochs, MD, Study Chair — Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Technische Universität München, Klinikum rechts der Isar, Department of Anesthesiology, Munich, Bavaria, Germany